CLINICAL TRIAL: NCT00542464
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation Safety, Pharmacodynamics, and Pharmacokinetics Study of Intravenous Imprime PGG™ Injection in Healthy Adult Subjects
Brief Title: Multiple-Dose, Dose-Escalation Safety, Pharmacodynamics, and Pharmacokinetics Study of Imprime PGG™ Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BIOBG-CL-002
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: Healthy
Keywords: Safety in Healthy Adult Subjects
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Placebo Comparator): 1.0 mg/kg Imprime PGG administered daily over 1 hr for 7 consecutive days
  Interventions: Biological: Imprime PGG TM for Injection
- Cohort 2 (Placebo Comparator): 2.0 mg/kg Imprime PGG administered daily over 1 hr for 7 consecutive days
  Interventions: Biological: Imprime PGG TM for Injection
- Cohort 3 (Placebo Comparator): 4.0 mg/kg Imprime PGG administered daily over 2 hr for 7 consecutive days
  Interventions: Biological: Imprime PGG TM for Injection

INTERVENTIONS:
Biological: Imprime PGG TM for Injection — Doses of 1.0 mg/kg-4.0 mg/kg of Imprime PGG administered over 1-2 hr for 7 consecutive days

SUMMARY:
The study is a Phase Ib, randomized, double-blind, placebo-controlled, multiple-dose (7 day), dose-escalation study assessing the safety, pharmacodynamics, and pharmacokinetics of intravenous Imprime PGG™ Injection in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 to 45 years, inclusive
2. Have a body weight of 45 to 125 kg, inclusive, and a body mass index less than or equal to 30 kg/m2
3. If female, be non-pregnant and non-nursing, and if pre-menopausal, have a negative serum pregnancy test confirmed prior to enrollment and practicing at least two methods of birth control
4. Be healthy as determined by the investigator on the basis of medical history, physical examination, electrocardiogram, and clinical laboratory test results
5. Have the ability to understand the requirements of the study, provide written informed consent, and agree to abide by the study restrictions and to return for the required assessments
6. Have provided written authorization for use and disclosure of protected health information

Exclusion Criteria:

1. Have a known hypersensitivity to baker's yeast
2. Have a history of tobacco use within 3 months of first day of screening
3. Be a known or suspected abuser of alcohol or other drugs/substances of abuse at anytime
4. Have an active yeast infection
5. Have a positive hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) test conducted as part of screening
6. Except as otherwise indicated, have taken any prescription medication within 30 days of the last day of screening (Day -1) or over-the-counter medication, herbal preparation, or vitamins within 7 days of the last day of screening (Day -1); the following medications are exempted from this criterion: acetaminophen [maximum 3 g/day], female hormone replacement therapy, and oral contraceptives
7. Have participated in an investigational drug study within 30 days or five half lives (whichever is longer) of the last day of screening (Day -1) or have ever participated in a study with Imprime PGG or Betafectin
8. Have donated or lost more than a unit of blood within 30 days of the last day of screening (Day -1)
9. Have any clinical condition that, in the opinion of the principal investigator, warrants exclusion from the study from a scientific, procedural, or safety perspective

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of 7 consecutive daily i.v. doses of Imprime PGG versus placebo when administered to healthy adult subjects by assessing the frequency, type, and severity of treatment-emergent adverse events (AE). | Prospective

SECONDARY OUTCOMES:
-To determine the pharmacodynamics of 7 consecutive daily intravenous doses of Imprime PGG by assessing the number of subjects who experience a 15% or more increase from baseline in the percentage of neutrophils with primed complement receptor (CR3). | Prospective
-To derive the pharmacokinetic profile of 7 consecutive daily intravenous doses of Imprime PGG when administered to healthy adult subjects by assessing the plasma concentration of Imprime PGG versus time profiles. | Prospective